CLINICAL TRIAL: NCT02332031
Title: An Open-label Study in Healthy Male Subjects to Assess the Effect of Hyperthyroidism Mimicked by Oral Dosing of Levothyroxine on the Pharmacokinetics of Sorafenib
Brief Title: Sorafenib Drug Drug Interaction Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 17436; 2014-001907-36 (EudraCT Number)
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Drug Interactions
Keywords: Sorafenib, levothyroxine, drug interaction, pharmacokinetics, healthy volunteer
MeSH Terms: interventions — Sorafenib; Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Nexavar, BAY43-9006) & Levothyroxine (Experimental): Sorafenib be administrated without and with levothyroxine orally
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Levothyroxine

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Single dose of 400 mg orally on Period 1 Day 1 and Period 2 Day 11
Drug: Levothyroxine — Single dose of 300 mcq orally from Period 2 Day 1 to Period 2 Day 14

SUMMARY:
To evaluate the effect of levothyroxine on the absorption, distribution, metabolization and elimination of sorafenib and safety in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 (inclusive) and 45 years (inclusive) at the first screening visit.
* Body mass index (BMI) between 18.5 (inclusive) to 30.0 kg / m² (inclusive) with body weight ≥ 65kg.
* Normal thyroid function indicated by thyroid examination to include total and free T3 (Triiodothyronine) , T4 (total and free Thyroxine, levothyroxine), TSH (Thyroid stimulating hormone), anti-TSH-receptor (anti-TSHR) antibody, anti-thyroperoxidase (anti-TPO) antibody, anti-thyroglobulin antibody (anti-ATA) as well as thyroid ultrasound.

Exclusion Criteria:

* History of clinically significant metabolic, renal, hepatic, or central nervous system disorder such as seizure, psychosis and sleep disorders.
* History of cardiovascular diseases including arrhythmia, hypertension, ischemia, etc.
* Known or suspected cardiovascular disease including potential risk of atrioventricular (AV) block, arrhythmia, etc. with or without a formal cardiologist consultation.
* Subjects who had received iodine containing contrast medium within 2 months before first study drug administration.
* Use of systemic or topical medicines or substances which might affect the study drug(s) must be avoided

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve from zero to infinity after single (first) dose (AUC) of sorafenib | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose

SECONDARY OUTCOMES:
AUC from time 0 to the last data point > LLOQ (AUC(0-tlast))of Sorafenib and metabolite M-2 | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of Sorafenib and metabolite M-2 | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Time to reach Cmax (in case of two identical Cmax values, the first tmax will be used) (Tmax Sorafenib) and metabolite M-2 | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Half-life associated with the terminal slope (t1/2) of Sorafenib and metabolite M-2 | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Apparent volume of distribution at steady state after extravascular administration (Vss/F) of Sorafenib | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Total body clearance of Sorafenib calculated after extravascular administration (CL/F) | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
AUC of metabolite M-2 | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Metabolite to parent AUC(0-tlast) ratios | Period 1 Day 1 and Period 2 Day 11: Predose and at 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 h post-dose
Number of participants with adverse events as a measure of safety and tolerability | Up to 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany